CLINICAL TRIAL: NCT00444691
Title: Sensitivity of Echography in Arthritis
Acronym: SEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Association de Recherche Clinique en Rhumatologie (Other)
Collaborators: RCTs (Industry)
Responsible Party: Professor Maxime DOUGADOS, Association de Recherche Clinique en Rhumatologie
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ARCR 2007/01; 2006-A00658-43
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Rheumatoid Arthritis
Keywords: synovitis score; sensitivity to change; clinical examination; ultra-sonography
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Tomography Scanners, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ultra-sonography — o The ultrasonographic evaluation was performed on 38 joints: the 28 joints included in DAS28 (e.g. shoulderx2, elbowx2, wristx2, metacarpo-phalangeal (MCP)x10, proximal inter phalangeal (PIP)x10, kneex2) and also the metatarso-phalangeal (MTPx10). Systematic multiplanar gray-scale (mode B) and Power Doppler examination was carried out with commercially available real-time scanners using multi-frequency linear transducers (7-12 MHz).
  The ultrasonographic evaluation was performed at baseline and 1, 2, 3, and 4 months after baseline.
  Other Names: scanners:; ESAOTE Technos MPX; TOSHIBA APLIO; ESAOTE MyLab; PHILIPS HD11; BK Mini Focus.

SUMMARY:
It has been reported recently that the detection of synovitis by ultrasonography was more sensitive than clinical examination (Wakefield et al. Ann Rheum Dis).

An OMERACT and EULAR working party recently produced guidelines on the best way to record and score quantitatively synovitis of the small joints of the hands and feet (Wakefield R, D'Agostino MA).

It has also been presumed recently that ultrasonography was more sensitive to changes than clinical examination after anti-TNF treatment (Ref. Taylor et al). If this better sensitivity to change were to be confirmed, ultrasonography would be preferred to clinical examination in studies evaluating new treatments.

In everyday practice, better intrinsic validity of the evaluation of synovitis by ultrasonography would lead to widespread use of this technique in the diagnosis and treatment of rheumatoid arthritis patients.

Objective of this study is to compare the sensitivity to change in synovitis score according to the monitoring method used (clinical examination versus ultrasonography).

DETAILED DESCRIPTION:
This is a multicenter, (10 French centers and 1 Belgian center), prospective (4-month patients' follow-up) interventional study in 120 patients with rheumatoid arthritis justifying anti-TNF treatment.

The overall duration of the study will be 8 months composed of a 4-month inclusion period and a 4-month follow-up period for each patient. Moreover, X-ray evaluations of hands and feet will be performed 2 years from the beginning of the study in order to assess the changes in structural damage.

During the patients' participation, 6 visits are planned: an inclusion visit then, a follow-up visit at 1, 2 and 3 months from the inclusion visit, and a final evaluation visit at 4 months from the inclusion visit. At each visit, synovitis will be evaluated using both methods: clinical examination and ultrasonography. For a same patient, clinical evaluation of synovitis will have to be performed - during the entire study - by the same rheumatologist and the ultrasonographic evaluation will have to be performed by the same ultrasonographist (different from the rheumatologist) and always using the same ultrasonograph.

Finally, patients will be performed anterior X-rays of hands and feet two years from the beginning of the study whatever the ongoing RA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis meeting ACR criteria.
* Justifying anti-TNF alpha treatment (switch or first administration).
* To have at least 6 synovitis at the clinical examination necessary for the DAS evaluation
* To accept to participate in this study (informed consent signed).

Exclusion Criteria:

* Minor patients.
* Pregnancy.
* Breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
joint score evaluated by clinical examination | baseline and 1, 2, 3 and 4 months after baseline
joint score evaluated by ultra-sonography | baseline and 1, 2, 3 and 4 months after baseline

SECONDARY OUTCOMES:
DAS28 Synovial index | baseline and 1, 2, 3 and 4 months after baseline
ACR Synovial index (66 sites) | baseline and 1, 2, 3 and 4 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Maxime DOUGADOS, Professor, Principal Investigator — ARCR
Locations (10):
- CHU-Brugmann, Brussels, Belgium
- France (9):
  - Hôpital Ambroise Paré, Boulogne
  - CHU de la Cavale Blanche, Brest
  - CHU Côte de Nacre, Caen
  - CHU A. Michallon, Grenoble
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Cochin, Paris
  - Hôpital de la Pitié, Paris
  - CHU de RENNES - Hôpital Sud, Rennes
  - CHU Nancy-Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Cheung PP, Mari K, Devauchelle-Pensec V, Jousse-Joulin S, D'Agostino MA, Chales G, Gaudin P, Mariette X, Saraux A, Dougados M. Predictive value of tender joints compared to synovitis for structural damage in rheumatoid arthritis. RMD Open. 2016 Mar 17;2(1):e000205. doi: 10.1136/rmdopen-2015-000205. eCollection 2016. PMID 27042336